CLINICAL TRIAL: NCT03628690
Title: A Post-Market Study of BandGrip in Traumatic Wound Closure Compared to Suture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BandGrip (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol: ERM-001, Version 01
Record Dates: First submitted 2018-07-18; First posted 2018-08-14 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Laceration of Skin
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Intervention Model Description: 2:1 randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- BandGrip (Experimental): Topical skin closure device
  Interventions: Device: BandGrip
- Standard Suture (Active Comparator): Standard sutures will be used for wound closure
  Interventions: Device: Suture

INTERVENTIONS:
Device: BandGrip — Topical skin closure device
  Arms: BandGrip
Device: Suture — Wound closure
  Arms: Standard Suture

SUMMARY:
an unbalanced (2:1) randomized study comparing two methods of traumatic skin closure in an ER setting: BandGrip vs suture

DETAILED DESCRIPTION:
Up to 45 subjects at up to 2 study sites who present to the ER for treatment of a skin laceration will be consented and randomized to treatment with suture or BandGrip. Subjects will be followed for 30 days post treatment to assess cosmetic quality of wound healing, evidence of adverse events related to closure method, and speed and completeness of wound closure and removal of closure devices.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female age 18-65.
* Subject presents to emergency room with at least one skin laceration that is assessed as requiring a suture closure on the trunk or extremities (excluding hands and feet).
* The length of the laceration is less than or equal to 1.5 inches.
* Subject is otherwise in good general health in the opinion of the investigator.
* Subject must be willing to follow instructions for wound care provided by investigator and refrain from picking at the treatment device, applying topical medications to the wound, and swimming or soaking in a tub until BandGrip or the sutures are removed.
* Subject agrees to return for follow-up evaluations.
* Subject (or guardian) is able to comprehend and give informed consent for participation in this study.

Exclusion Criteria:

* Significant multiple trauma (merely multiple wounds are allowed).
* The wound involves a lower limb with critical limb ischemia.
* Concurrent acute infection requiring intravenous or oral antibiotics.
* Bleeding, coagulation and or clotting disorders.
* Subject is on dialysis.
* Inflammatory and or allergic diseases or conditions of the skin: for example, psoriasis, eczema or dermatitis.
* History of drug abuse.
* Chronic use of oral steroids or immunosuppressants.
* Known personal or family history of keloid or hypertrophic scarring.
* History of abnormal wound healing.
* Burst stellate lacerations due to a crush or hard blow.
* Animal or human bite or scratch.
* Wound is in the head, hands or feet or in a high skin tension area or across an area of increased skin tension on a joint.
* Investigator objects to a patient's involvement in the study protocol.
* Known allergy to components to BandGrip or suture material.
* Known cognitive or psychiatric disorder.
* Wound requiring debridement of devitalized or contaminated tissue.
* Wound at site of active rash/skin lesion making evaluation difficult.
* Previously treated wound or has failed to heal.
* Puncture wound.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Complete wound closure | 30 days post treatment
  defined as continuous approximation of skin margins without need for reintervention .

SECONDARY OUTCOMES:
Wound comesis | 10 and 30 days post closure
  a 100mm visual analog scale (with 100 representing complete satisfaction with comesis) assessing wound cosmesis using the Comesis Visual Analog Scale.
Pain/discomfort | index procedure and 10 days post closure
  The subject will complete a 100mm visual analog scale with 100 representing worst pain level.
Infection | 10 and 30 days post closure
  incidence of clinical infection requiring antibiotic treatment.
Subject satisfaction | 30 days post closure
  subjects will complete a 100mm VAS (with 100 representing complete satisfaction) to evaluate their overall assessment of their scar,
Physician satisfaction | index procedure
  a 100mm VAS ( with 100mm representing complete satisfaction) to evaluate the overall ease of wound closure.
Time to wound closure and device removal | index procedure and 10 days post wound closure
  Time to closure and removal of closure device
Subject Satisfaction | 30 days post closure
  indication of subject preference for method of sound closure
Wound Evaluation | 10 and 30 days post wound closure
  assessment of the quality of wound healing by the physician.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Donohoe, Study Director — BandGrip
Locations (1):
- University of Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No